CLINICAL TRIAL: NCT01309009
Title: Double-blind, Randomised, Placebo-controlled, Parallel Group Pilot Study to Evaluate the Efficacy and Safety of Oral Administration of Nepadutant in Infant Colic Babies Not Responder to Conventional Treatments
Brief Title: Preliminary Efficacy and Safety Study of Oral Nepadutant in Infant With Colic Not Responding to Conventional Treatment
Acronym: nocry-a
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIC-05 (NOCRY-a)
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Infantile Colic
Keywords: Infantile Colic; Tachykinin antagonist; Nepadutant
MeSH Terms: conditions — Colic | interventions — MEN 11420

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nepadutant High Dose (Experimental)
  Interventions: Drug: Nepadutant oral solution
- Nepadutant Low Dose (Experimental)
  Interventions: Drug: Nepadutant oral solution
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching Nepadutant oral solution

INTERVENTIONS:
Drug: Nepadutant oral solution — Oral administration once daily for 7 days
  Arms: Nepadutant Low Dose
Drug: Placebo matching Nepadutant oral solution — Oral administration once daily for 7 days
  Arms: Placebo
Drug: Nepadutant oral solution — Oral administration once daily for 7 days
  Arms: Nepadutant High Dose

SUMMARY:
This phase IIa study is designed as a multi-centre, single country, randomised, double-blind, placebo controlled study in three parallel groups, with the aim to evaluate the efficacy and safety of Nepadutant given at two oral doses once daily for seven days in comparison to placebo in the treatment of infantile colic.

DETAILED DESCRIPTION:
Infant colic is a functional gastrointestinal disorders which affects up to the 30% of the infant population; it is primarily characterised by excessive inconsolable crying starting without any apparent cause and lasting for several hours per day.

Current non pharmacological interventions (e.g. message, restriction in maternal diet in breast-feeding infants) and pharmacological treatments (simethicone, antimuscarinic drugs) are largely unsatisfactory.

In animal models, Nepadutant reverse the exaggerated intestinal motility and sensitivity, induced by different stimuli, without producing inhibitory effects on these functions at baseline, suggesting that Nepadutant could have a therapeutic effect with no interference on physiological gastrointestinal transit.

This phase IIa study is designed to evaluate the efficacy of Nepadutant paediatric oral solution given once daily at two doses in comparison to placebo.

The experimental clinical phase encompasses the following periods:

* Screening period (no study medication) to be done 7 to 4 days prior to randomisation
* Treatment period, lasting seven days with once daily administration
* Post treatment period, lasting seven days A safety follow-up visit will be performed approximately 1 month after the first administered dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants with diagnosis of infant colic according to the following modified Wessel criterion "paroxysm of irritability, fussing or crying that start and stop without obvious cause for >3h/day, >3 days/week for one week"
* Age ≥ 6 weeks and < 4 months
* No adequate response to conventional pharmacological or non-pharmacological treatment alternatives for infant colic
* Infants exclusively breast-fed.
* Normal growth
* Willingness to refrain from use of antimuscarinic drugs, simethicone, dimethicone or antiacids during the study period

Exclusion Criteria:

* Clinical evidence of allergies or other diseases which may cause crying and/or fussiness or may interfere with absorption or clearance of the drug.
* Suspect of gastroesophageal reflux disease (GERD)
* Formula fed or mixed fed infants.

Ages: 6 Weeks to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Absolute change of the mean daily crying and fussing time for three consecutive days while on treatment versus baseline. | one week

SECONDARY OUTCOMES:
Percentage of 'responder' babies at the end of treatment period. | one week
Absolute change in the overall parental judgment after the first dose of treatment, at the end of treatment, and after treatment discontinuation versus baseline. | ten days
Safety and tolerability will be assessed in terms of frequency and severity of AEs as well as frequency of clinically significant changes in physical examination and lab test. | up to four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Lionetti, MD, Study Chair — Servizio di Gastroenterologia dell'Azienda Ospdedaliero - Universitaria Anna Meyer di Firenze